CLINICAL TRIAL: NCT06295588
Title: Minimizing Fatigue and Inflammation in Survivors of Cancer: A Pilot Randomized Clinical Trial of the Seaweed Supplement Fucoidan
Brief Title: Clinical Trial of the Seaweed Supplement Fucoidan in Survivors of Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeremy J McGuire, Research Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009135; T32CA102618 (NIH)
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Fatigue; Inflammation
Keywords: cancer-related fatigue
MeSH Terms: conditions — Fatigue; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fucoidan (Experimental): They will receive 4 grams daily of fucoidan extracted from F. Vesiculosus for 8 weeks.
  Interventions: Drug: Fucoidan extracted from F. Vesiculosus
- Usual Care (Active Comparator): They will receive usual care for 8 weeks followed by 4 grams daily of fucoidan extracted from U. Pinnatifida for 8 weeks.
  Interventions: Drug: Fucoidan extracted from U. Pinnatifida

INTERVENTIONS:
Drug: Fucoidan extracted from F. Vesiculosus — 4 g daily
  Arms: Fucoidan
Drug: Fucoidan extracted from U. Pinnatifida — 4 g daily
  Arms: Usual Care

SUMMARY:
To determine the feasibility of an 8-week fucoidan supplement intervention for patients with fatigue post-cancer treatment and assess changes in fatigue, frailty, and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of cancer
* Age 18 or older
* Speak and understand English
* Have completed surgery, radiation, and/or systemic intravenous anticancer therapy (e.g., chemotherapy, targeted therapy, immunotherapy) ≤10 years prior to enrollment.
* Have a baseline level of fatigue, as determined by reporting a score of 4 or higher for the question, "In the last week, how bad was your worst fatigue on a scale from 0-10?"
* Be willing to commit to the fucoidan supplement dosing and delivery method, to complete evaluation instruments, and to attend all study visits.
* Completed Informed Consent

Exclusion Criteria:

* Current warfarin or other anti-coagulation medication use.
* Current use of supplements that contain fucoidan
* Any allergy to fucoidan
* Be diagnosed with a major psychiatric illness requiring hospitalization within the last year.
* Be diagnosed with dementia.
* Be pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
percentage of participants who are randomized to the study out of all participants approached | 8 weeks
percentage of participants who start the intervention who go on to complete the 8-week or 16-week intervention | 16 weeks
percentage of participants who take at least 80% of the fucoidan pills during the study | 8 weeks

SECONDARY OUTCOMES:
mean change in Brief Fatigue Inventory | baseline to 16 weeks
  The Brief Fatigue Inventory is a 9-item questionnaire that ranges from 0 to 10 with higher scores indicating a worse outcome.
mean change in plasma viscosity in blood | baseline to 16 weeks
mean change in erythrocyte sedimentation rate in blood | baseline to 16 weeks
mean change in thyroid stimulating hormone in blood | baseline to 16 weeks
mean change in C-reactive protein in blood | baseline to 16 weeks
mean change in leptin in blood | baseline to 16 weeks
mean change in D Dimer in blood | baseline to 16 weeks
mean change in TNF alpha in blood | baseline to 16 weeks
mean change in neopterin in blood | baseline to 16 weeks
mean change in lactase dehydrogenase in blood | baseline to 16 weeks
mean change in procalcitonin in blood | baseline to 16 weeks
mean change in frailty using a modified Fried's Frailty questionnaire | baseline to 16 weeks
  The modified Fried's Frailty questionnaire measures self-reported slowness, weakness, weight loss, physical activity and fatigue. The total score of the questionnaire ranges from 1 to 5 with higher numbers indicating worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No